CLINICAL TRIAL: NCT03491943
Title: Midline Versus Paramedian Approaches for Ultrasound-assisted Spinal Anesthesia: a Randomized Controlled Trial
Brief Title: Midline vs. Paramedian Approaches for US-assisted Spinal Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin-Tae Kim, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: H-1803-060-928
Record Dates: First submitted 2018-04-02; First posted 2018-04-09 (Actual); Last update posted 2019-12-23 (Actual); Status verified 2019-12

CONDITIONS: Anesthesia, Spinal; Ultrasonography

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Midline group (Experimental): Preprocedural ultrasound-assisted midline approach of spinal anesthesia will be performed. 0.5% heavy bupivacaine will be injected to intrathecal space for spinal anesthesia.
  Interventions: Procedure: ultrasound-assisted midline approach
- Paramedian group (Active Comparator): Preprocedural ultrasound-assisted paramedian approach of spinal anesthesia will be performed. 0.5% heavy bupivacaine will be injected to intrathecal space for spinal anesthesia.
  Interventions: Procedure: ultrasound-assisted paramedian approach

INTERVENTIONS:
Procedure: ultrasound-assisted midline approach — A preprocedural ultrasound scanning will be done, and skin marking will be made. The needle entry point and insertion angle will be determined based on ultrasound scanning. Spinal anesthesia will be performed via midline approach.
  Arms: Midline group
Procedure: ultrasound-assisted paramedian approach — A preprocedural ultrasound scanning will be done, and skin marking will be made. The needle entry point and insertion angle will be determined based on ultrasound scanning. Spinal anesthesia will be performed via paramedian approach.
  Arms: Paramedian group

SUMMARY:
Ultrasound has emerged as an useful tool for neuraxial blockade. The aim of this study is to compare the efficacy and safety between the midline approach and paramedian approach for ultrasound-assisted spinal anesthesia in adult patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients scheduled to undergoing elective orthopedic surgery under spinal anesthesia, with ASA physical status classification I, II, III

Exclusion Criteria:

* Patients with contraindication to spinal anesthesia (coagulopathy, local infection, allergy to local anesthetic)
* Patients with morbid cardiac diseases
* Pregnancy
* Patients with previous history of lumbar spinal surgery
* Patients with anatomical abnormality of lumbar spine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2018-04-27 (Actual); Primary Completion 2018-10-08 (Actual); Study Completion 2018-10-09 (Actual)

PRIMARY OUTCOMES:
the number of needle passes | Intraoperative (from the first insertion of needle to patient's skin, until the completion of spinal anesthetic injection)
  the number of forward advancements of the spinal needle in a given interspinous space, i.e., withdrawal and redirection of spinal needle without exiting the skin

SECONDARY OUTCOMES:
Number of spinal needle insertion attempts | Intraoperative (from the first insertion of needle to patient's skin, until the completion of spinal anesthetic injection)
  the number of times the spinal needle was withdrawn from the skin and reinserted
Time for identifying landmarks | intraoperative (time taken for establish the landmark, from start of US scanning to completion of scanning
  time from placement of the ultrasound probe on the skin to the completion of markings.
Time taken for performing spinal anesthetic | Intraoperative (from insertion of the needle to the completion of injection)
  time from needle insertion to the completion of injection
dermatome level of sensory block | 20 minutes after the completion of spinal anesthetic injection
  thoracic dermatome level of sensory block assessed by loss of cold sensation tested with 2% chlorhexidine swab
Incidence of radicular pain, paraesthesia, and blood tapping in the spinal needle | Intraoperative (from the first insertion of needle, until the completion of spinal anesthetic injection)
  Incidence of radicular pain, paraesthesia, and blood tapping in the spinal needle during the spinal anesthesia procedure
Periprocedural pain | Patients will be asked immediately after the completion of spinal anesthesia
  11-point verbal rating scale (0=no pain, 10=most pain imaginable)
Periprocedural discomfort score | Patients will be asked immediately after the completion of spinal anesthesia
  11-point verbal rating scale (0=no discomfort, 10=most discomfort imaginable)
Patient satisfaction score of spinal anesthesia procedure | Patients will be asked immediately after the completion of spinal anesthesia
  11-point verbal rating scale (0=very unsatisfied, 10=very satisfied)

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Tae Kim, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kallidaikurichi Srinivasan K, Iohom G, Loughnane F, Lee PJ. Conventional Landmark-Guided Midline Versus Preprocedure Ultrasound-Guided Paramedian Techniques in Spinal Anesthesia. Anesth Analg. 2015 Oct;121(4):1089-1096. doi: 10.1213/ANE.0000000000000911. PMID 26270115
- [Derived] Park SK, Cheun H, Kim YW, Bae J, Yoo S, Kim WH, Lim YJ, Kim JT. Ultrasound-assisted spinal anesthesia: A randomized comparison between midline and paramedian approaches. J Clin Anesth. 2022 Sep;80:110823. doi: 10.1016/j.jclinane.2022.110823. Epub 2022 Apr 11. PMID 35421679